CLINICAL TRIAL: NCT02666599
Title: Per-operating Use of a Probe for Detection of β+
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, John O. Prior, Chief of Nuclear Medicine Department, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 363/11
Record Dates: First submitted 2016-01-24; First posted 2016-01-28 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Neoplasms
Keywords: F-18-FDG; neoplasm; probe; positron; diagnosis; surgery; radioguided surgery
MeSH Terms: conditions — Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-FDG PET/CT (Experimental): 18F-FDG radiotracer All patients will undergo a 18F-FDG PET/CT and a surgery with probe detection of β+''
  Interventions: Radiation: 18F-FDG PET/CT

INTERVENTIONS:
Radiation: 18F-FDG PET/CT — A 18F-FDG PET/CT will be done. A dose of 19 µSv/MBq will be received by the patient. Surgery will be conducted within 3 hours after the I.V. injection of 18F-FDG according to the standard procedure applied in the visceral surgery department. During the surgery, emission of β+ from the lesion (s) seen durint the PET/CT will be detected with the probe.
  Resected pieces will be analysed histologically.

SUMMARY:
The objective of the study is to evaluate the sensibility of the probe Forimtech to detect β+ emission in vivo in humans and its usefulness during elective surgical procedure Hypothesis:The probe Forimtech is able to allow per-surgery detection of tumoral lesions sensible to 18F-FDG and to help in the realization of guided biopsies, minimally invasive surgery or complement of resection of tumors.

The β+ emission detected by the probe Forimtech is correlated to the emission γ detected by the 18F-FDG.PET/CT

DETAILED DESCRIPTION:
Patients with a malignant neoplasic lesion known or suspected for which a surgery is planned will be presented with the protocol. If inclusion/exclusion criteria are fulfilled all the procedures will be planned. A 18F-FDG PET/CT will be done. Surgery will be conducted within 3 hours after the I.V. injection of 18F-FDG according to the standard procedure applied in the visceral surgery department. During the surgery, emission of β+ from the lesion (s) seen during the PET/CT will be detected with the probe.

Resected pieces will be analysed histologically.

ELIGIBILITY:
Inclusion Criteria:

* Age < 80 years old;
* Karnofsky index ≥80% ;
* Informed consent signed
* Patients with an indication of thoracic, visceral, or ENT surgery with the aim of a diagnostic biopsy, of an invasive minimal treatment, or an initial or complementary resection

Exclusion Criteria:

* Pregnancy
* Enable to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Sensibility of the probe β+ for detection per-surgery of hypermetabolic tumoral lesions | day 0
  Topography and intensity of detection by the probe of emission of β+ by the lesion(s)
  • Intensity of emission of β+ by the non specific background and the adjacent structures

SECONDARY OUTCOMES:
PET/CT imaging results | day 0
  * 18F-FDG PET imaging: SUVmax of the lesion(s), SUVmean of the lesion(s), ratio SUVmax / SUVbackground
  * CT imaging: Topography of / the lesion(s), size of / the lesion(s), distance with the surrounding organs
Sensibility of the probe β+ for detection per-surgery of hypermetabolic tumoral lesions | within 10 days after study procedure
  Change in every primary interpretation criterion corresponding to the parameters of detection found during the operation will be studied and compared with the analysis of the parameters of the histology (gold standard) through an analysis ROC. They will be also studied compared with the analysis of the parameters PET/ CT
.Comparison of AUC of the imaging methods | within 10 days after study procedure
  A comparison of the AUC will be realized to determine the superiority of a method compared with the other one, by a non parametric test comparing AUC, ROC curves respectively

CONTACTS AND LOCATIONS:
Overall Officials: John O Prior, PhD MD, Principal Investigator — Lausanne University Hospitals
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Vaus, Switzerland

IPD SHARING:
Plan to Share IPD: No